CLINICAL TRIAL: NCT01521780
Title: A Clinical Study to Characterize Baseline Biomarker Variability in Participants With Hepatocellular Carcinoma for Utilization of Target Engagement and Pharmacodynamic Biomarkers in Future Phase I Trials
Brief Title: Characterization of Baseline Biomarker Variability in Participants With Hepatocellular Carcinoma (MK-0000-215)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-215
Record Dates: First submitted 2011-12-16; First posted 2012-01-31 (Estimated); Results first posted 2013-10-28 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; MRI; pharmacogenomics; beta-catenin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imaging (Experimental): Magnetic resonance imaging (MRI) of HCC tumor.
  Interventions: Procedure: MRI; Procedure: Blood Samples
- Pathology (Experimental): Pathology samples from surgical resection of HCC tumor and adjacent liver.
  Interventions: Procedure: Pathology; Procedure: Blood Samples
- Imaging/Pathology (Experimental): MRI of HCC tumor, followed by pathology samples from surgical resection of HCC tumor and adjacent liver.
  Interventions: Procedure: MRI; Procedure: Pathology; Procedure: Blood Samples

INTERVENTIONS:
Procedure: MRI — Participants undergo volumetric & diffusion weighted (DW) MRI. Participants are scanned twice, with an intervening fifteen minute walk between the scans.
  Arms: Imaging; Imaging/Pathology
Procedure: Pathology — Participants who are undergoing surgical resection of HCC per their standard of care treatment, will submit tumor samples for biomarker analysis.
  Arms: Imaging/Pathology; Pathology
Procedure: Blood Samples — Blood is collected from participants during screening Visit 1 - 24.5 ml. During Visit 3, blood samples totaling 22 ml, are collected at least 6-18 hours post-resection, and every other day up to a week until discharge. At follow up Visit 4, 5.5 ml of blood is collected.
  Arms: Imaging/Pathology; Pathology
Procedure: Blood Samples — Blood is collected from participants during screening Visit 1 - 24.5 ml, and follow up Visit 4 - 5.5 ml.
  Arms: Imaging

SUMMARY:
The purpose of this study is to characterize the baseline variability of a panel of tissue (tumor and adjacent) and blood-based biomarkers obtained from participants with hepatocellular carcinoma (HCC). The primary hypothesis is that the upper bound of the 80% Confidence Interval of log beta-catenin protein or messenger RNA (mRNA) expression from one core needle biopsy (CNB) equivalent is =< 0.65.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCC.
* Candidate for surgical resection or has no contraindications to MRI procedures.

Exclusion Criteria:

* Prior loco-regional treatment of tumor, unless there is untreated tumor present representing a distinct untreated nodule.
* Confirmed or suspected diagnosis of fibrolamellar HCC, mixed HCC/cholangiocarcinoma or metastatic tumor.
* Had a liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Imaging: Magnetic resonance imaging (MRI) of Hepatocellular carcinoma (HCC) tumor.
Period: Overall Study
Arm/Group | Imaging | Pathology | Imaging/Pathology
Started | 9 | 1 | 2
Completed | 9 | 1 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants who enrolled in the study
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Expression Levels of Beta-catenin mRNA From Core Needle Biopsy (CNB) Equivalents of Resected HCC.
Description: Resected tumors were fixed with formalin in paraffin embedded (FFPE) blocks, which were used to prepare multiple serial slide sections. The sections were to be analyzed for beta-catenin messenger RNA (mRNA) by quantitative reverse transcription polymerase chain reaction (qRT-PCR).
Time Frame: Visit 3, approximately 7 days after screening Visit 1.
Population: Due to early termination of the study, the low number of samples were not assayed and efficacy analyses were not performed.
Arm/Group | Imaging | Pathology | Imaging/Pathology
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Expression Levels of Beta-catenin Protein From Core Needle Biopsy (CNB) Equivalents of Resected HCC.
Description: Resected tumors were fixed in FFPE blocks, which were used to prepare multiple serial slide sections. The sections were to be analyzed for beta-catenin protein by automated image analysis.
Time Frame: Visit 3, approximately 7 days after screening Visit 1.
Population: as for outcome 1
Arm/Group | Imaging | Pathology | Imaging/Pathology
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Tumor Volumes From Repeated MRI Measurements of HCC.
Description: Two volumetric MRI and diffusion weighted (DW) MRI scans were performed without contrast on each participant. The two scans were separated by 10 to 15 minutes, and each scan was read by a separate reader to determine the volume of each tumor. The mean of log tumor volume is presented, based on tumors as observation units.
Time Frame: Visit 2, approximately 7 days after screening Visit 1.
Population: Eleven participants underwent MRI and DW MRI scans and only ten of their tumors were deemed measurable by both readers for analysis. Participants in both the Imaging and Imaging/Pathology treatment groups were combined for this analysis, whereas participants in the Pathology only treatment group were not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: log cm^3
Units Other Than Participants: Tumors
Groups:
- Imaging and Imaging/Pathology: Magnetic resonance imaging (MRI) of HCC tumor.
Arm/Group | Imaging and Imaging/Pathology
Number analyzed (Participants) | 11
Number analyzed (Tumors) | 10
log cm^3 | 3.38 (0.235)
Statistical Analysis 1: Comparison: Imaging and Imaging/Pathology; Test type: Superiority or Other; Within subject coefficient of variation = 0.0803, 90% CI 1-sided [upper limit 0.1163]

4. Secondary Outcome: Median Apparent Diffusion Coefficient (Median ADC) of Tumors From Repeated MRI Measurements of HCC.
Description: Two volumetric MRI and diffusion weighted (DW) MRI scans were performed without contrast on each participant. The two scans were separated by 10 to 15 minutes, and each scan was read by a separate reader to derive a Median ADC for each tumor. The mean of the Median ADCs is presented based on tumours as observation units.
Time Frame: Visit 2, approximately 7 days after screening Visit 1.
Population: Eleven participants underwent MRI and DW MRI scans and only eight of their tumors were deemed measurable by both readers for analysis. Participants in both the Imaging and Imaging/Pathology treatment groups were combined for this analysis, whereas participants in the Pathology only treatment group were not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: um^2/s
Units Other Than Participants: Tumors
Arm/Group | Imaging and Imaging/Pathology
Number analyzed (Participants) | 11
Number analyzed (Tumors) | 8
um^2/s | 1340.56 (64.45)
Statistical Analysis 1: Comparison: Imaging and Imaging/Pathology; Test type: Superiority or Other; Within subject coefficient of variation = 0.0555, 90% CI 1-sided [upper limit 0.0733]

5. Secondary Outcome: Expression Levels of Beta-catenin mRNA From CNB Equivalents of Liver Adjacent to HCC.
Description: Tissues adjacent to resected tumors were fixed in FFPE blocks, which were used to prepare multiple serial slide sections. The sections were to be analyzed for beta-catenin mRNA by qRT-PCR.
Time Frame: Visit 3, approximately 7 days after screening Visit 1.
Population: as for outcome 1
Arm/Group | Imaging | Pathology | Imaging/Pathology
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Expression Levels of Beta-catenin Protein From CNB Equivalents of Liver Adjacent to HCC.
Description: Tissues adjacent to resected tumors were fixed in FFPE blocks, which were used to prepare multiple serial slide sections. The sections were to be analyzed for beta-catenin protein by automated image analysis.
Time Frame: Visit 3, approximately 7 days after screening Visit 1.
Population: as for outcome 1
Arm/Group | Imaging | Pathology | Imaging/Pathology
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Expression Levels of Low Density Lipoprotein Receptor (LDL-R) in Resected HCC and Adjacent Liver From Whole Tissue Sections.
Description: Resected tumors and adjacent tissues were fixed in FFPE blocks, which were used to prepare multiple serial slide sections. The sections were to be analyzed for LDL-R protein by automated image analysis.
Time Frame: Visit 3, approximately 7 days after screening Visit 1.
Population: as for outcome 1
Arm/Group | Imaging | Pathology | Imaging/Pathology
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Imaging | Pathology | Imaging/Pathology
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/9 | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.